CLINICAL TRIAL: NCT04361812
Title: A Multicenter, Randomized, Double-blind, Parallel Controlled，Single-dose Phase I Study Comparing the Pharmacokinetic and Safety Similarities of Recombinant Anti IgE Humanized Monoclonal Antibody (HS632) With Omalizumab a in Healthy Subjects
Brief Title: Comparison of Pharmacokinetics and Safety of HS632 and Xolair® With a Single Injection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company R&D Strategy Adjustment
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS632-I
Record Dates: First submitted 2020-04-14; First posted 2020-04-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Similarity of Pharmacokinetics and Safety
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS632 (Experimental): HS632 150mg for a single subcutaneous injection
  Interventions: Drug: HS632
- Omalizumab (Xolair®) (Active Comparator): Omalizumab 150mg for a single subcutaneous injection
  Interventions: Drug: Omalizumab (Xolair®)

INTERVENTIONS:
Drug: HS632 — Subcutaneous injection of HS632
  Other Names: Recombinant anti IgE humanized monoclonal antibody 150mg
  Arms: HS632
Drug: Omalizumab (Xolair®) — Subcutaneous injection of Omalizumab Xolair®)
  Other Names: Omalizumab 150mg
  Arms: Omalizumab (Xolair®)

SUMMARY:
To evaluate the bioequivalence of HS632 and Omalizumab (Xolair®) in a single subcutaneous administration in healthy subjects.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel controlled，single-dose phase I study to compare the pharmacokinetic and safety similarities of recombinant anti IgE humanized monoclonal antibody (HS632) With omalizumab a in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1.Signing the informed consent and being able to complete the test according to the plan;
* 2.Age ≥ 18 and ≤ 40 (subject to the date of signing the informed consent), male;
* 3.The body mass index (BMI) is between 20and6 kg / m2 (including 20 kg / m2 and 26 kg / m2), and the body weight is between 50-75 kg (including 50 kg and 75 kg);
* 4.The subject (including the partner) has no plan of pregnancy from the date of signing informed consent to 6 months after the administration of the experimental drug and is willing to use effective contraceptive methods, such as abstinence, oral contraceptives, iUDs or double barrier methods (e.g., condom plus diaphragm)

Exclusion Criteria:

* 1.Patients with mental, respiratory, cardiovascular, digestive, urinary, reproductive, skeletal and motor, blood, endocrine, nervous and other system diseases, or patients with any previous immune diseases;
* 2.Patients with severe bleeding factors affecting venous blood collection
* 3.Skin diseases or other diseases affecting subcutaneous injection;
* 4. Patients with upper respiratory tract infection or other acute infection in the 2 weeks prior to screening;
* 5.Patients with history of malignant tumor;
* 6.Those who have undergone surgery within two months before signing the informed consent;
* 7.Drinking more than 14 units of alcohol per week (14 bottles of 360 ml beer or 630ml of 40% spirits or 2100ml of wine) within 6 months before screening, or those with positive results of alcohol breath test;
* 8.Those who have used soft drugs (e.g., marijuana) within 3 months prior to signing the informed consent or hard drugs (e.g., cocaine, phencyclidine, etc.) within 1 year prior to the trial； those who have positive drug abuse test results (morphine, methamphetamine, ketamine, MDMA, tetrahydrocannabinolic acid, cocaine);
* 9. Those who are addicted to smoking or smoke more than 5 cigarettes per day on average in the 3 months before signing the informed consent; or those who have positive nicotine results;
* 10.Those who have a history of drug or food allergy, or who have special requirements for diet and cannot abide by the unified diet or specific allergy history (asthma, urticaria, eczema dermatitis, etc.); those who have allergic rhinitis, or are known to be allergic to any component of the test drug or latex (contained in the syringe needle cover);
* 11.Those who drinking too much tea, coffee and / or caffeinated beverages (more than 8 cups, 1 cup = 250 ml) every day;
* 12. Those who have received any drug treatment (including prescription drugs, over-the-counter drugs, biological products, Traditional Chinese medicine, vitamins, dietary supplements, etc.) and health care products within 14 days before signing the informed consent;
* 13. Traditional Chinese medicine (except proprietary Chinese Medicine) and health care products are planned to be used during the test;
* 14. Have a blood donation history within 3 months before signing the informed consent, or plan to donate blood during the trial;
* 15. Those who plan to accept any biological drugs within 3 months after the administration of the test drug or those who plan to accept monoclonal antibody drugs within 9 months;
* 16. Those who plan to donate sperm within 6 months after the administration of the test drug;
* 17. Those who plan to undergo (including cosmetic surgery, dental surgery and oral surgery) during the trial period;
* 18. Those who plan to take part in strenuous exercise during the experiment, including physical contact exercise or collision exercise;
* 19. Participants in other clinical trials within 3 months before signing the informed consent;
* 20. Vaccinated within 6 months before signing the informed consent;
* 21. In the screening period or baseline period, the researchers think that the physical examination and laboratory examination of the subjects have clinical significance abnormalities; or the following indicators exceed the following standards: the rate of pulse in awake state is less than 50 times / min or more than 100 times / min, the systolic pressure in sitting position is equal to or more than 140 mmHg or the diastolic pressure is more than 90 mmHg, and the ear temperature is more than 37.5 ℃; any one of eosinophil, neutrophil, platelet is beyond the normal range; eGFR is less than 90 mL / min / 1.73m2 (estimated by MDRD formula of kidney disease diet improvement test, see Annex I);
* 22. Patients with clinically significant ECG abnormalities in screening or baseline period, or with QTcF ≥ 450 ms, or with a history of clinically significant ECG abnormalities in the past;
* 23. The results of chest X-rayor chest CT examination or B-ultrasonic examination are clinically significant abnormalities according to the judgment of the researcher;
* 24.Any one of HIV antibody, HBsAg, HBeAg, HBcAg, HCV antibody and Treponema pallidum antibody is positive;
* 25. The researchers think those who are considered by the investigator unsuitable for the trail or who may not be able to complete the trial for other reasons is not suitable to be enrolled or may not be able to complete the experiment for other reasons;
* 26. Employees or relatives of researchers, research centers, sponsors and contract research organizations.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
AUC(0 -∞) of single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Area Under the concentration-time Curve from time zero to infinity of single subcutaneous administration of HS632 and Xolair in healthy subjects
Cmax of single subcutaneous administration of HS632 and Xolair in healthy subjects Peak plasma concentration (Cmax) after single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Maximum serum concentration (Cmax) of HS632 and Xolair in healthy subjects Peak plasma concentration (Cmax) after single subcutaneous administration of HS632 and Xolair in healthy subjects

SECONDARY OUTCOMES:
AUC (0 - t) of HS632 and Xolair in single subcutaneous administration in healthy subjects | 13weeks
  Area under the plasma concentration versus time curve (AUC) from 0 to the last selected time point, i.e. 2184h after the injection
2.Tmax of single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Time to Cmax (Tmax) of single subcutaneous administration of HS632 and Xolair in healthy subjects
3.CLt/F of single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Total clearance corrected by bioavailability (CLt/F) of single subcutaneous administration of HS632 and Xolair in healthy subjects
Half-life (T1/2) of single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Half-life (T1/2) of single subcutaneous administration of HS632 and Xolair in healthy subjects
Vd/F of single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Apparent volume of distribution corrected by bioavailability (Vd/F) of single subcutaneous administration of HS632 and Xolair in healthy subjects
Incidence of Treatment-Emergent Adverse Events[Safety] | 13weeks
  Incidence of Treatment-Emergent Adverse Events [Safety] of distribution corrected by bioavailability (Vd/F) of single subcutaneous administration of HS632 and Xolair in healthy subjects
Immunogenicity of single subcutaneous administration of HS632 and Xolair in healthy subjects | 13weeks
  Anti drug antibody（ADA）of single subcutaneous administration of HS632 and Xolair in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Dr. Pharm, Principal Investigator — Huashan Hospital; Xiaojie Wu, Dr. Pharm, Principal Investigator — Huashan Hospital
Locations (1):
- Anhui Peng, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No